CLINICAL TRIAL: NCT03128060
Title: Expanding Access to Home-Based Palliative Care Through Primary Care Medical Groups
Brief Title: Expanding Access to Home-Based Palliative Care
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study enrollment was terminated due to inability to recruit participants
Sponsor: University of Southern California (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Susan Enguidanos, Associate Professor of Gerontology, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PCORI-1234
Record Dates: First submitted 2017-04-16; First posted 2017-04-25 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Cancer; Congestive Heart Failure; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Palliative Care (Experimental): Home-based palliative care features home visits by an interdisciplinary PC team (physician, nurse, social worker, and chaplain) that provides pain and symptom management, psychosocial support, advance care planning, disease management education, spiritual and grief counseling, and other services as needed.
  Interventions: Other: Home-based palliative care
- Enhanced Usual Care (Active Comparator): Enhanced usual care refers to: 1) usual primary care provided by a primary care physician who has been offered special training in the core elements of palliative care; 2) case management services; and 3) provider support through palliative care consultation.
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Other: Home-based palliative care — The HBPC model consists of home visits by an interdisciplinary primary palliative care team (a physician, nurse, social worker, and chaplain). This team provides pain and symptom management, psychosocial support, advance care planning, spiritual counseling, grief counseling, and other services to meet patient and caregiver needs. Within the first week of a patient's enrollment, team members separately visit the patient at home to assess his/her needs as well as the needs of his/her caregiver. Following the patient's initial assessment, subsequent home visits are based on the patient's and caregiver's needs. At a minimum, a core team member visits the patient at home once per week. Additionally, a 24/7 helpline provides access to nurse counseling and after-hours home visits as needed. As a patient's health declines and he/she becomes eligible for hospice care, HBPC clinicians will refer the patient to hospice.
  Other Names: Home-based primary palliative care
  Arms: Home-based Palliative Care
Other: Enhanced usual care — Usual primary care consists of: 1) appointment-based access to primary care providers (PCPs) as requested by the patient; 2) case management services; and 3) provider support through palliative care consultation. These PCPs provide family/internal medicine services as well as access to specialist care. They also offer disease case management and pain and symptom management.
  These usual care services are enhanced through training in palliative care provided to PCPs. The training addresses core elements of palliative care, specifically these 6 topics: a palliative care overview; strategies for improving patient-provider communications; instruction in ACP; instruction in managing patients' pain and symptoms; care coordination; and preventing medical crises.
  Arms: Enhanced Usual Care

SUMMARY:
This study will test the effectiveness of integrating an evidence-based model of home-based palliative (HBPC) within primary care clinics on patient and caregiver outcomes. The investigators will conduct a randomized controlled trial, randomizing 1,155 seriously ill patients (and approximately 884 family caregivers) who receive primary care from 30-40 regional accountable care organizations (ACOs) in California to one of two study groups: HBPC or enhanced usual care (EUC). Follow-up data will be collected via telephone surveys with patients at 1- and 2-months and with caregivers at 1- and 2-months, and, as appropriate, following the death of the patient.

DETAILED DESCRIPTION:
Background and Significance

Patients with serious illness from cancer, heart failure (HF), and chronic obstructive pulmonary disease (COPD) often receive poor quality of care, resulting in unmitigated pain and related symptoms, unmet psychosocial needs, and significant caregiver burden. Palliative care, a patient-centered approach that provides pain and symptom management and psychosocial and spiritual support, has strong evidence for improved outcomes for these seriously ill patients. Palliative care differs from hospice in that it is offered early in the illness course and in conjunction with other therapies intended to prolong life. Most palliative care programs are hospital-based; few offer care at home, where patients spend the most time and require the most support.

Study Aims

This study will test the effectiveness of integrating an evidence-based model of home-based palliative (HBPC) within primary care clinics on patient and caregiver outcomes. The investigators will conduct a randomized controlled trial, randomizing 1,155 seriously ill patients (and approximately 884 family caregivers) who receive primary care from 30-40 regional accountable care organizations (ACOs) in California to one of two study groups: HBPC or enhanced usual care (EUC). Follow-up data will be collected via telephone surveys with patients at 1- and 2-months and with caregivers at 1- and 2-months, and, as appropriate, following the death of the patient.

The study's specific aims are:

* Specific Aim 1: Determine differences in improvement on measures of physical and psychological well-being between patients receiving HBPC and patients receiving enhanced usual care (EUC).
* Specific Aim 2: Determine differences in survival time between patients receiving HBPC and patients receiving EUC.
* Specific Aim 3: Determine differences in number of emergency department (ED) visits and hospital admissions between patients receiving HBPC and patients receiving EUC.
* Specific Aim 4: Determine differences in improvement on patient-provider communication between patients receiving HBPC and patients receiving EUC.
* Specific Aim 5: Determine differences in improvement on psychosocial outcomes between caregivers of patients receiving HBPC and caregivers of patients receiving EUC.

Study Description

Study Population. The study will enroll 1,155 patients and approximately 883 caregivers from primary care medical groups operating under ACO contracts with Blue Shield of California (Blue Shield), the study's insurance partner. About 75% of patients will be age 65 or older; about 55% will be female. About 45% of patients will be ethnic minority members, predominantly of Hispanic decent.

Comparators. The study will compare outcomes from two groups: patients who receive EUC (with usual care enhanced by: 1) provider training in palliative care; 2) case management for EUC patients; and 3) provider support through palliative care consultation) and patients who receive HBPC provided by an HBPC team. HBPC features home visits by an interdisciplinary PC team (physician, nurse, social worker, and chaplain) that provides pain and symptom management, psychosocial support, advance care planning, disease management education, spiritual and grief counseling, and other services as needed.

Outcomes. Primary outcomes are change in patient pain, symptoms, depression, and anxiety. These measures will be collected via patient self-report at baseline and at one- and two-months following enrollment. Change in survival, ED visits, and hospital episodes (including length of stay, when applicable) also are primary outcomes that will be collected from the electronic medical record (EMR). These data will be collected following patient death or at study's end. Secondary patient outcomes are peace, patient-physician communication, and hope.Secondary caregiver outcomes are change in caregiver depression, anxiety, burden, and patient-physician communication, with these assessments all collected at baseline and one- and two-months following enrollment. Caregiver's experience of patient death will be collected one month following patient death, when applicable.

Analytic Methods. Investigation of the main effect of HBPC and EUC on outcomes will be conducted at each follow-up and then on the longitudinal trend. Baseline outcome measures will be treated as covariates to control for potential baseline differences. Repeated measures analyses will be used to investigate the longitudinal effects of program conditions on outcome measures. Sub-analyses will examine outcome differences by patient age, diagnosis, and race.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older;
2. diagnosis of HF, COPD, or advanced cancer;
3. one or more hospitalizations or ED visits in the previous year;
4. an Australia-Modified Karnofsky Performance Scale score of 70% or less; and
5. English- or Spanish-speaking.

Exclusion Criteria:

1. is receiving hospice care;
2. has end-stage renal disease; and/or
3. lives in a nursing home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-08-19 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Enguidanos, Ph.D., Principal Investigator — USC Davis School of Gerontology
Locations (1):
- USC Davis School of Gerontology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Enguidanos S, Rahman A, Lomeli S. A Tale of Two Trials: A Comparative Case Study of Successful versus Terminated Home-Based Palliative Care Trials. J Palliat Med. 2022 Dec;25(12):1767-1773. doi: 10.1089/jpm.2022.0065. Epub 2022 Jun 8. PMID 35675655
- [Derived] Enguidanos S, Rahman A. Early Termination of a Palliative Care Trial: Perspectives of Multiple Stakeholders on Barriers to Palliative Care and Research. J Palliat Med. 2022 Jan;25(1):54-59. doi: 10.1089/jpm.2021.0234. Epub 2021 Jun 30. PMID 34191594
- [Derived] Enguidanos S, Rahman A, Fields T, Mack W, Brumley R, Rabow M, Mert M. Expanding Access to Home-Based Palliative Care: A Randomized Controlled Trial Protocol. J Palliat Med. 2019 Sep;22(S1):58-65. doi: 10.1089/jpm.2019.0147. PMID 31486727

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Target sample size: 1,155 patients, 884 caregivers
Groups:
- Home-based Palliative Care - Patients; Home-based Palliative Care - Caregivers: Home-based palliative care features home visits by an interdisciplinary PC team (physician, nurse, social worker, and chaplain) that provides pain and symptom management, psychosocial support, advance care planning, disease management education, spiritual and grief counseling, and other services as needed.
  Home-based palliative care: The HBPC model consists of home visits by an interdisciplinary primary palliative care team (a physician, nurse, social worker, and chaplain). This team provides pain and symptom management, psychosocial support, advance care planning, spiritual counseling, grief counseling, and other services to meet patient and caregiver needs. Within the first week of a patient's enrollment, team members separately visit the patient at home to assess his/her needs as well as the needs of his/her caregiver. Following the patient's initial assessment, subsequent home visits are based on the patient's and caregiver's needs. At a minimum, a core team member visits the patient at home once per week. Additionally, a 24/7 helpline provides access to nurse counseling and after-hours home visits as needed. As a patient's health declines and he/she becomes eligible for hospice care, HBPC clinicians will refer the patient to hospice.
- Enhanced Usual Care - Patients; Enhanced Usual Care - Caregivers: Enhanced usual care refers to: 1) usual primary care provided by a primary care physician who has been offered special training in the core elements of palliative care; 2) case management services; and 3) provider support through palliative care consultation.
  Enhanced usual care: Usual primary care consists of: 1) appointment-based access to primary care providers (PCPs) as requested by the patient; 2) case management services; and 3) provider support through palliative care consultation. These PCPs provide family/internal medicine services as well as access to specialist care. They also offer disease case management and pain and symptom management.
  These usual care services are enhanced through training in palliative care provided to PCPs. The training addresses core elements of palliative care, specifically these 6 topics: a palliative care overview; strategies for improving patient-provider communications; instruction in ACP; instruction in managing patients' pain and symptoms; care coordination; and preventing medical crises.
Period: Overall Study
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
Started | 13 | 15 | 3 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 13 | 15 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers | Total
Number analyzed (Participants) | 13 | 15 | 3 | 4 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.1 (12.6) | 64.2 (12.6) | 48.0 (11.8) | 57.0 (7.9) | 66.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 10 | 2 | 3 | 20
  Male | 8 | 5 | 1 | 1 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 0 | 2
  Not Hispanic or Latino | 11 | 15 | 2 | 4 | 32
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 12 | 11 | 2 | 4 | 29
  More than one race | 1 | 2 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1
Marital Status [Count of Participants; unit: Participants]
  Married | 10 | 9 | 3 | 4 | 26
  Single | 1 | 2 | 0 | 0 | 3
  Widowed | 1 | 3 | 0 | 0 | 4
  Divorced | 1 | 1 | 0 | 0 | 2
Religion [Count of Participants; unit: Participants] — Caregiver's religion was not collected. Population: Not collected for caregivers
  Participants
    number analyzed (Participants) | 13 | 15 | 0 | 0 | 28
    Agnostic | 0 | 1 | 0 | 0 | 1
    Catholic (Christian) | 5 | 1 | 0 | 0 | 6
    Christian (other) | 7 | 8 | 0 | 0 | 15
    None / Atheist | 1 | 5 | 0 | 0 | 6
Income [Count of Participants; unit: Participants]
  Less than $20,000 | 5 | 0 | 1 | 1 | 7
  $20,000 - $ 199,999 | 8 | 13 | 2 | 3 | 26
  $200,000 or more | 0 | 1 | 0 | 0 | 1
  Unknown | 0 | 1 | 0 | 0 | 1
Education [Count of Participants; unit: Participants]
  Less than high school | 1 | 1 | 0 | 0 | 2
  High school graduate | 3 | 1 | 1 | 1 | 6
  Some college | 4 | 5 | 1 | 2 | 12
  College graduate | 1 | 5 | 1 | 1 | 8
  Post-graduate school | 4 | 2 | 0 | 0 | 6
  Unknown | 0 | 1 | 0 | 0 | 1
Hospital Anxiety and Depression Scale (HADS_PT_CG) [Mean (Standard Deviation); unit: score on a scale] | 16.8 (6.0) | 18.6 (4.5) | 6.0 (8.7) | 10.8 (7.1) | 17.8 (5.2)
Patient Health Questionnaire (PT) [Mean (Standard Deviation); unit: score on a scale] — Caregiver's Patient Health Questionnaire was not collected. Population: Not collected for caregivers
  score on a scale
    number analyzed (Participants) | 13 | 15 | 0 | 0 | 28
    (all) | 11.0 (5.2) | 12.9 (5.1) |  |  | 12.0 (5.2)
Edmonton Symptom Assessment Scale [Mean (Standard Deviation); unit: units on a scale] — Caregiver's Edmonton Symptom Assessment Scale was not collected. Population: Not collected for caregivers
  units on a scale
    number analyzed (Participants) | 13 | 15 | 0 | 0 | 28
    (all) | 37.7 (14.4) | 32.1 (16.4) |  |  | 34.7 (15.5)
Herth Hope Index (PT) [Mean (Standard Deviation); unit: units on a scale] — Caregiver's Herth Hope Index was not collected. Population: Not collected for caregivers
  units on a scale
    number analyzed (Participants) | 13 | 15 | 0 | 0 | 28
    (all) | 38.2 (5.1) | 35.0 (5.5) |  |  | 36.5 (5.5)
Assessment of Peace (PT) [Mean (Standard Deviation); unit: units on a scale] — Caregiver's Assessment of Peace was not collected. Population: 1 missing in HBPC group
  units on a scale
    number analyzed (Participants) | 12 | 15 | 0 | 0 | 27
    (all) | 3.8 (0.8) | 2.9 (1.0) |  |  | 3.33 (1.0)
Consultation Care Measure (PT_CG) [Mean (Standard Deviation); unit: units on a scale] | 48.2 (10.9) | 56.6 (13.1) | 40.0 (21.2) | 52.5 (9.7) | 52.7 (12.7)

OUTCOME MEASURES:

1. Primary Outcome: Edmonton Symptom Assessment Survey for Patients
Description: The Edmonton Symptom Assessment Survey for patients is a brief and reliable self-report assessment that measures the frequency and intensity of a variety of physical and psychological symptoms. Response scores range from 0 (no pain/symptoms) to 90 (highest pain symptoms) based on responses scored from 0 (no pain/symptoms) to 10 (highest pain/symptoms) on 9 items. Note: our data represents the composite score of the 9 items.
Time Frame: 1-month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 35.2 (12.5) | 28.1 (10.6)

2. Primary Outcome: Hospital Anxiety and Depression Scale (HADS) for Patients
Description: The Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire that measures anxiety and depression using a 4-point Likert scale. The assessment consists of 14 patient-reported items, with seven questions reflecting anxiety (HADS-A) and seven reflecting depression (HADS-D). The total score for each subscale ranges from 0 to 21, and the total score is the sum of the two subscale scores. Low scores indicate normal responses while high scores are abnormal (0-7 = Normal, 8-10 = Borderline abnormal, 11-21 = Abnormal).
Time Frame: 1-month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 15.9 (6.9) | 14.4 (2.9)

3. Secondary Outcome: Patient Health Questionnaire-9 (PHQ-9) for Patients
Description: The Patient Health Questionnaire-9 is a 9-item assessment to diagnose depression, with each item scores from 0 (not at all) to 3 (nearly every day). It is based on the nine DSM-IV criteria for depression. Scores range from a minimum of 0 to a maximum of 27. Low scores indicate no depression, while high scores indicate depression. For example, a score of 15 or greater is considered major depression, 20 or more is severe major depression.
Time Frame: 1-months following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 10.8 (5.4) | 8.7 (4.5)

4. Secondary Outcome: Rating of Being at Peace Among Patients
Description: This is a 1-item probe that assesses an individual's feeling of being at peace. On a scale of 1 to 5, with 1 being "Not at all at peace," and 5 being "Completely at peace". High scores indicate better outcomes. Scores range from a minimum of 1 (worse outcome) to a maximum of 5 (best outcome).
Time Frame: 1-month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 4.0 (1.2) | 3.2 (0.8)

5. Secondary Outcome: Hearth Hope Index for Patients
Description: The Hearth Hope Index is a 12-item scale is used to assess hope as it relates to a person's ability to cope with medical illness, loss, and related psychosocial stressors. The scale for each question ranges from 1 (strongly disagree) to 4 (strongly agree), with the exception of items 3 and 6, which are reverse-coded. Possible scores range from 12 to 48, with higher scores indicating higher level of hope (positive outcome).
Time Frame: 1-month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 37.7 (2.8) | 37.3 (3.6)

6. Secondary Outcome: Consultation Care Measure (CCM) for Patients
Description: The Consultation Care Measure (CCM) is a patient-reported assessment evaluates patient-physician relationships, including communication, approach to the problem, and interest in the patient's life. WThis measure includes 20 likert scale questions for with response ranging from 1 to 4 for each (1 = very strongly agree... 4 = Neutral/disagree). The total score ranges from 20 to 80 and the lower score is the better score.
Time Frame: At 1 months following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients
Number analyzed (Participants) | 9 | 10
score on a scale | 43.9 (10.8) | 56.7 (13.0)

7. Secondary Outcome: Zarit Burden: Short (ZBI) Interview Among Caregivers
Description: The Zarit Burden Interview: Short (ZBI) is a 12-item instrument that has been used with caregivers for a wide range of patients, including those with chronic illnesses. Total score range is 0 to 48, with higher scores indicating higher burden. Interpretation of score: 0-10=no to mild burden; 10-20= mild to moderate burden; and > 20= high burden.
Time Frame: At 1 month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
Number analyzed (Participants) | 2 | 1
score on a scale | 7.5 (10.6) | 17

8. Secondary Outcome: Caregiver's Experience of Death Rating on Family Assessment of Treatment at End of Life- Short Form (FATE-S), When Applicable.
Description: FATE-S scores are expressed as a percentage of valid responses for which families provided the best possible response; higher percentages reflect better experience of care.
Time Frame: Two months following the death of a patient
Population: * There were no patient deaths during the study period.
Arm/Group | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Hospital Anxiety and Depression Scale (HADS) for Caregivers
Description: as for outcome 2
Time Frame: At 1 month following baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
Number analyzed (Participants) | 2 | 1
score on a scale | 6.5 (9.2) | 0

10. Secondary Outcome: Consultation Care Measure (CCM) for Caregivers
Description: This caregiver-reported assessment evaluates patient-physician relationships, including communication, approach to the problem, and interest in the patient's life. The Consultation Care Measure (CCM)assessment evaluates patient-physician relationships, including communication, approach to the problem, and interest in the patient's life. This measure includes 20 likert scale questions for with response ranging from 1 to 4 for each (1 = very strongly agree... 4 = Neutral/disagree). The total score ranges from 20 to 80 and the lower score is the better score.
Time Frame: At 1- month following baseline
Population: Only two caregivers reported follow-up CCM, both of them are in HBPC group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
Number analyzed (Participants) | 2 | 0
score on a scale | 32.5 (23.3) |

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Home-based Palliative Care - Patients | Enhanced Usual Care - Patients | Home-based Palliative Care - Caregivers | Enhanced Usual Care - Caregivers
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/13 | 1/15 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/13 | 0/15 | 0/3 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Home-based Palliative Care - Patients (N=13) | Enhanced Usual Care - Patients (N=15) | Home-based Palliative Care - Caregivers (N=3) | Enhanced Usual Care - Caregivers (N=4)
ER visit or hospitalization (General disorders) | 2 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Home-based Palliative Care - Patients (N=13) | Enhanced Usual Care - Patients (N=15) | Home-based Palliative Care - Caregivers (N=3) | Enhanced Usual Care - Caregivers (N=4)
Severe pain (General disorders) | 2 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
After 18 months of significant enrollment challenges, largely based on our health insurance company providing palliative care to everyone who qualified and subsequent challenges in obtaining patient referrals to the study, we elected to terminate the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/60/NCT03128060/Prot_000.pdf